CLINICAL TRIAL: NCT04587882
Title: Virtual AppLication-supported ENvironment To INcrease Exercise During Cardiac Rehabilitation Study
Acronym: VALENTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Corewell Health West (Other)
Responsible Party: Principal Investigator, Brahmajee K Nallamothu, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00162365
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Heart Diseases; Cardiovascular Diseases
Keywords: Cardiac rehabilitation
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: A prospective, randomized-controlled trial where the primary purpose is secondary prevention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): Participants will be provided with a smartwatch, have access to activity tracking and goal setting through the VALENTINE app, receive micro-randomized, contextually tailored notifications, and receive weekly activity summaries via email, which will be provided to participants and to their exercise physiologist while enrolled in cardiac rehabilitation.
  Interventions: Behavioral: Telehealth
- Control (Active Comparator): Participants will continue to receive usual care and a smartwatch but without access to the micro-randomized notifications or weekly activity summaries.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Telehealth — Participants will receive weekly activity summaries and tailored notifications about their activity and goal setting behaviors.
  Arms: Telehealth
Behavioral: Control — Participants will get usual care and wear a smartwatch.
  Arms: Control

SUMMARY:
The researchers are trying to determine whether a smartwatch and a mobile application, which together deliver activity and goal setting notifications, can increase activity levels for patients enrolled in cardiac rehabilitation.

DETAILED DESCRIPTION:
The VALENTINE Cardiac Rehabilitation Study will evaluate a digital intervention to supplement cardiac rehabilitation for low- and moderate risk patients, integrating a mobile application with physiologic and contextual information from wearables to provide incremental support to patients. The study will be performed in conjunction with planned home-, hybrid-, or center-based cardiac rehabilitation at Michigan Medicine. Participants will be randomized to the control or telehealth group. Both groups will receive a smartwatch and usual care. Participants in the telehealth arm will additionally (1) have access to activity tracking and goal setting through the VALENTINE app; (2) receive micro-randomized, contextually tailored notifications, and (3) receive weekly activity summaries via email, which will also be provided to their exercise physiologist while enrolled in cardiac rehabilitation. Contextually tailored notifications will be one of two types: walking and exercise notifications. Walking notifications are designed to encourage participants to be active though at lower than their target heart rate zone. Participants will receive 1 notification per day, on average, at one of four times. Notifications will be randomized on four dimensions of context. Exercise notifications are designed to encourage participants to exercise within their target heart rate zone. Notifications will be delivered each evening at a time of the participant's choosing. Participants will have a 50% probability of receiving a notification each evening. Notifications will be randomized on two dimensions of context. Participants will be followed for 6-months. Participants in both arms will be asked to complete a 6-minute walk test at baseline, 3-months, and 6-months using their mobile phone and smartwatch. They will additionally complete general and disease-specific quality-of-life questionnaires at baseline and at 6-months.

To account for potential measurement error between devices, for primary and secondary analyses, we will perform regression analysis to jointly test the null hypothesis H0: B0(F) = B0(A) = 0 for change between baseline and 6 months where (F) and (A) refer to Fitbit and Apple watches respectively. A secondary analysis will subsequently be performed to determine whether to reject the individual null hypotheses for each of the two devices. For all statistical analyses, the level of significance will be set at p <0.05.

ELIGIBILITY:
Inclusion criteria:

1. Must be a patient within the Michigan Medicine clinical system with data available in the electronic health record after January 1, 2013. Spectrum Health patients may participate if they have a Michigan Medicine MRN and data is available through connected electronic health records.
2. Age > 18 and < 75
3. Owns an Android or iPhone with study supported operating software.
4. Understands English to enable informed consent, completion of study-related surveys, and compliance with study notifications.
5. Enrolled in cardiac rehabilitation within the past 8-weeks based on one of the following indications (listed below) and has completed at least 2 cardiac rehabilitation sessions (includes orientation session; to remain in the study, participants in the hybrid program must complete at least one additional exercise session for a minimum of 2 center-based rehabilitation sessions):

   * Coronary artery disease (including acute coronary syndromes and stable angina) following percutaneous coronary intervention (PCI)
   * Coronary artery disease following coronary artery bypass surgery (CABG)]
   * Valve repair or replacement (either surgical or percutaneous)
   * Coronary artery disease or an acute coronary syndrome not requiring revascularization

Exclusion criteria:

1. Orthopedic or neurological condition limiting ability to actively engage in exercise training session
2. Greater than mild cognitive impairment
3. Wrist too large to wear a smartwatch comfortably. This will be assessed by asking participants "If they have ever had difficulty wearing a watch in the past due to the band being too small."
4. Currently receiving palliative care and/or in hospice care
5. Severe valvular stenosis or regurgitation
6. Unrevascularized left main coronary artery disease (> 50% obstruction on angiography) or proximal left anterior descending disease (>70% obstruction on angiography).
7. Exercise-induced ventricular tachycardia
8. Cardiac arrest within the prior 6 months
9. New York Heart Association (NYHA) class III or IV heart failure
10. Pulmonary arterial hypertension treated with inhaled or intravenous pulmonary hypertension-specific therapy
11. Ejection fraction <40%
12. Determined to be unsafe for participation in this program to augment cardiac rehabilitation as assessed by a clinical nurse or investigative team.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | Baseline, 6-months
  6-minute walk distance is determined by the 6-minute walk test recorded using a mobile phone paired with a smartwach and recorded in meters.

SECONDARY OUTCOMES:
Change in average step count | Baseline, 6-months
  Change in average step count as determined by smartwatch. Baseline average is the average step count from the first 7 days of wearing the smartwatch. The 6-month average step count is the daily average step count over one week at 6-months.

OTHER OUTCOMES:
Proximal outcome for activity notifications. | 1-hour after an activity notification, up to 6-months.
  The proximal outcome for activity notifications will be average step count 1-hour after a notification measured by smartwatch.
Proximal outcome for exercise notifications. | The day after an exercise notification, up to 6-months.
  The proximal outcome for exercise notifications will be exercise minutes the day after a notification, defined as the number of "fairly active" and "very active" minutes on smartwatch.
All-cause mortality and Cardiovascular mortality | 6-months
  The event numbers will be added together
All-cause mortality and Cardiovascular mortality | 12-months
  The event numbers will be added together
Cardiovascular hospitalizations | 6-months
Cardiovascular hospitalizations | 12-months
Change in 6-minute walk distance | Baseline, 3-months
  6-minute walk distance is determined by the 6-minute walk test recorded using a mobile phone paired with a smartwach and recorded in meters.
Change in 6-minute walk distance, subgroup analysis | Baseline and 6-months
  6-minute walk distance is determined by the 6-minute walk test recorded using a mobile phone paired with a smartwach and recorded in meters. Outcome measures will be stratified by type of cardiac rehabilitation, duration of cardiac rehabilitation, age, gender, baseline walk distance, and comfort with digital technology.
Change in average step count, subgroup analysis | Baseline and 6-months
  Change in average step count as determined by smartwatch. Baseline average is the average step count from the first 7 days of wearing the smartwatch. The 6-month average step count is the daily average step count over one week at 6-months. Outcome measures stratified by type of cardiac rehabilitation, age, gender, baseline walk distance, and comfort with digital technology.
Subgroup analyses of micro-randomized notifications by notification type | 6-months
  Subgroup analyses will be performed to determine which notification types are most effective based on the following features: Loss versus gain framework; Emoji versus no emoji in message; Message personalized with name versus no name ; Message includes hyperlink to study dashboard versus no hyperlink; Message encourages an activity versus anti-sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Brahmajee K Nallamothu, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golbus JR, Shi J, Gupta K, Stevens R, Jeganathan VSE, Luff E, Boyden T, Mukherjee B, Kohnstamm S, Taralunga V, Kheterpal V, Kheterpal S, Resnicow K, Murphy S, Dempsey W, Klasnja P, Nallamothu BK. Text Messages to Promote Physical Activity in Patients With Cardiovascular Disease: A Micro-Randomized Trial of a Just-In-Time Adaptive Intervention. Circ Cardiovasc Qual Outcomes. 2024 Jul;17(7):e010731. doi: 10.1161/CIRCOUTCOMES.123.010731. Epub 2024 Jun 18. PMID 38887953
- [Derived] Atluri N, Mishra SR, Anderson T, Stevens R, Edwards A, Luff E, Nallamothu BK, Golbus JR. Acceptability of a Text Message-Based Mobile Health Intervention to Promote Physical Activity in Cardiac Rehabilitation Enrollees: A Qualitative Substudy of Participant Perspectives. J Am Heart Assoc. 2024 Jan 16;13(2):e030807. doi: 10.1161/JAHA.123.030807. Epub 2024 Jan 16. PMID 38226512
- [Derived] Golbus JR, Gupta K, Stevens R, Jeganathan VS, Luff E, Boyden T, Mukherjee B, Klasnja P, Kheterpal S, Kohnstamm S, Nallamothu BK. Understanding Baseline Physical Activity in Cardiac Rehabilitation Enrollees Using Mobile Health Technologies. Circ Cardiovasc Qual Outcomes. 2022 Jul;15(7):e009182. doi: 10.1161/CIRCOUTCOMES.122.009182. Epub 2022 May 13. PMID 35559648
- [Derived] Jeganathan VS, Golbus JR, Gupta K, Luff E, Dempsey W, Boyden T, Rubenfire M, Mukherjee B, Klasnja P, Kheterpal S, Nallamothu BK. Virtual AppLication-supported Environment To INcrease Exercise (VALENTINE) during cardiac rehabilitation study: Rationale and design. Am Heart J. 2022 Jun;248:53-62. doi: 10.1016/j.ahj.2022.02.012. Epub 2022 Feb 27. PMID 35235834